CLINICAL TRIAL: NCT06683352
Title: A PHASE 1/2, RANDOMIZED, OBSERVER-BLINDED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF COMBINED VACCINE CANDIDATES AGAINST INFLUENZA AND COVID-19 IN HEALTHY INDIVIDUALS
Brief Title: A Study to Learn About Flu and COVID-19 Vaccine Responses in Healthy People
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C5261023
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Influenza,Human; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19 | interventions — COVID-19 Vaccines; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Arm A (Experimental): COVID-19 Vaccine (Dose 1) and Placebo
  Interventions: Biological: COVID-19 Vaccine; Other: Placebo
- Arm B (Experimental): COVID-19 Vaccine (Dose 2) and Placebo
  Interventions: Biological: COVID-19 Vaccine; Other: Placebo
- Arm C (Active Comparator): COVID-19 Vaccine (Dose 3) and Placebo
  Interventions: Biological: COVID-19 Vaccine; Other: Placebo
- Arm D (Experimental): Investigational Influenza Vaccine (Dose 1) and Placebo
  Interventions: Biological: Investigational Influenza Vaccine; Other: Placebo
- Arm E (Active Comparator): Licensed Influenza Vaccine 1 and COVID-19 Vaccine (Dose 3)
  Interventions: Biological: COVID-19 Vaccine; Biological: Licensed Influenza Vaccine 1
- Arm EE (Active Comparator): Licensed Influenza Vaccine 2 and COVID-19 Vaccine (Dose 3)
  Interventions: Biological: COVID-19 Vaccine; Biological: Licensed Influenza Vaccine 2
- Arm F (Experimental): Investigational Influenza Vaccine (Dose 2) and Placebo
  Interventions: Biological: Investigational Influenza Vaccine; Other: Placebo
- Arm G (Experimental): Influenza and COVID Combination Vaccine (Combination 1) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo
- Arm H (Experimental): Influenza and COVID Combination Vaccine (Combination 2) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo
- Arm I (Experimental): Influenza and COVID Combination Vaccine (Combination 3) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo
- Arm J (Experimental): Investigational Influenza Vaccine (Dose 3) and Placebo
  Interventions: Biological: Investigational Influenza Vaccine; Other: Placebo
- Arm K (Experimental): Influenza and COVID Combination Vaccine (Combination 4) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo
- Arm L (Experimental): Influenza and COVID Combination Vaccine (Combination 5) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo
- Arm M (Experimental): Influenza and COVID Combination Vaccine (Combination 6) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo
- Arm N (Experimental): Influenza and COVID Combination Vaccine (Combination 7) and Placebo
  Interventions: Combination Product: Influenza and COVID Combination Vaccine; Other: Placebo

INTERVENTIONS:
Biological: Investigational Influenza Vaccine — Investigational Influenza Vaccine
  Arms: Arm D; Arm F; Arm J
Biological: COVID-19 Vaccine — Pfizer-BioNTech COVID-19 Vaccine
  Arms: Arm A; Arm B; Arm C; Arm E; Arm EE
Combination Product: Influenza and COVID Combination Vaccine — Combined investigational influenza and Pfizer-BioNTech COVID-19 Vaccine
  Arms: Arm G; Arm H; Arm I; Arm K; Arm L; Arm M; Arm N
Biological: Licensed Influenza Vaccine 1 — Licensed Influenza Vaccine 1
  Arms: Arm E
Biological: Licensed Influenza Vaccine 2 — Licensed Influenza Vaccine 2
  Arms: Arm EE
Other: Placebo — Saline
  Arms: Arm A; Arm B; Arm C; Arm D; Arm F; Arm G; Arm H; Arm I; Arm J; Arm K; Arm L; Arm M; Arm N

SUMMARY:
This study is to learn about flu and COVID vaccines, either alone or when mixed together. Healthy people aged 18 or older can join. Participants will get one shot in each arm, either a flu or COVID vaccine, alone or mixed. The study lasts about 6 months, and participants need to visit the research site at least 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age or older
* Healthy participants who are determined by medical history, physical examination (if clinically required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Exclusion Criteria:

* Vaccination with any investigational or licensed 2024-2025 season formulation influenza or COVID-19 vaccine.
* Treated with antiviral therapies for influenza (eg, Tamiflu) within 180 days prior to Day 1

Please refer to the study contact for further eligibility details.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1353 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting prompted local reactions within 7 days following investigational product administration | Day 7
  Describe prompted local reactions following investigational product administration
Percentage of participants reporting prompted systemic events within 7 days following investigational product administration | Day 7
  Describe prompted systemic events following investigational product administration
Percentage of participants reporting adverse events (AEs) through 4 weeks following investigational product administration | 4 weeks after vaccination
  Describe AEs occurring through 4 weeks following administration of investigational product
Percentage of participants reporting serious adverse events (SAEs) through 6 months following investigational product administration | 6 months after vaccination
  Describe SAEs through 6 months following administration of investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Orange County Research Center, Lake Forest, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinical Research Professionals, Chesterfield, Missouri
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO-Screening and Recruitment Center, Springfield, Missouri
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - DM Clinical Research- Cyfair, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5261023